CLINICAL TRIAL: NCT00707603
Title: Understanding the Relationship Between Insulin Resistance and Chronic Hepatitis C Infection
Brief Title: Chronic Hepatitis C and Insulin Resistance
Status: Completed | Type: Observational
Sponsor: Garvan Institute of Medical Research (Other)
Responsible Party: Principal Investigator, Dr Jerry Greenfield, Head of Endocrinology Department St Vincent's Hospital Sydney, Garvan Institute of Medical Research
Other Study IDs: H04/126
Record Dates: First submitted 2008-06-29; First posted 2008-07-01 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C; Insulin Resistance
Keywords: Insulin resistance; Liver fat; Muscle fat; Abdominal fat; Cytokines
MeSH Terms: conditions — Hepatitis C; Insulin Resistance; Fatty Liver

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hepatitis C subjects: Due to start therapy for Hepatitis C
- Controls: Healthy males

SUMMARY:
Chronic hepatitis C (CHC) is among the commonest chronic infectious disease in Australia with >200,000 exposed persons. Amongst non-infectious chronic conditions- Type 2 diabetes, obesity and heart disease are extremely common. This study will examine the relationship between insulin resistance, fat deposition in the liver, muscle and abdomen, and liver injury due to CHC

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male
* Age: 25-55 years
* Chronic Hepatitis C (PCR positive) and fibrosis ≤ F2 (if liver biopsy done)
* Genotypes 1 or 3
* Due to commence antiviral therapy
* BMI < 30

Exclusion Criteria:

* Cirrhosis or F3 fibrosis on liver biopsy (if done)
* > 20 g ETOH per day
* Type 2 Diabetes (need an OGTT if fasting BGL> 5.7)
* Concurrent HIV
* Other cause of liver disease

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Hepatitis C patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance by euglycaemic hyperinsulinaemic clamp Liver fat, abdominal fat and muscle fat measures | 2 years

SECONDARY OUTCOMES:
insulin resistance post treatment of Hep C | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald Chisholm, MBBS, FRACP, Principal Investigator — Garvan Institute of Medical Research; Jacob George, MBBS, FRACP, Principal Investigator — Storr Liver Unit
Locations (2):
- Australia (2):
  - Garvan Institute Of Medical Research, Sydney, New South Wales
  - Storr Liver Unit, Sydney, New South Wales

REFERENCES:
- [Derived] Milner KL, van der Poorten D, Trenell M, Jenkins AB, Xu A, Smythe G, Dore GJ, Zekry A, Weltman M, Fragomeli V, George J, Chisholm DJ. Chronic hepatitis C is associated with peripheral rather than hepatic insulin resistance. Gastroenterology. 2010 Mar;138(3):932-41.e1-3. doi: 10.1053/j.gastro.2009.11.050. Epub 2009 Dec 4. PMID 19962985